CLINICAL TRIAL: NCT04621591
Title: Case Series With Saneso 3600 Gastroscope
Brief Title: Case Series With Saneso 360° Gastroscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saneso Inc. (Industry)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SAN360UGICL
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: EGD Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Saneso 360° gastroscope (Experimental): Subjects will have a clinically indicated per standard of care EGD procedure performed using the Saneso 360° gastroscope. Immediately thereafter Patients will then have an EGD procedure using a standard Gastroscope (Olympus GIF 180) performed by a second endoscopist.
  Interventions: Device: Saneso 360° gastroscope

INTERVENTIONS:
Device: Saneso 360° gastroscope — Subjects will have a clinically indicated per standard of care routine EGD procedure performed with the Saneso 360° gastroscope.

SUMMARY:
To confirm the procedural performance of the Saneso 360° gastroscope in Esophago-gastro-duodenoscopy (EGD) procedures.

DETAILED DESCRIPTION:
This study is a prospective, multicenter case series per standard of care EGD procedures using a nonsignificant risk Saneso 360° gastroscope. 20 cases will be included at up to five (5) clinical sites. Patients who meet all eligibility criteria will be included and will have a clinically indicated EGD procedure performed using the study device. Immediately thereafter, patients will have an EGD procedure using a standard Gastroscope (Olympus GIF180) by a second endoscopist. Enrolled subjects will be followed for 7 days after their procedure. If the procedure is not successful with the study device, the endoscopist will complete the procedure with a traditional gastroscope used at each facility.

ELIGIBILITY:
Inclusion Criteria:

* 18 -74 years of age
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.
* Scheduled for a clinically indicated routine EGD procedure
* ASA class 1-3.

Exclusion Criteria:

* Altered esophageal, gastric, or duodenal anatomy
* Pregnant women, children under 18 years of age, and adults over 75 years of age.
* Subjects for whom routine endoscopic procedures are contraindicated due to comorbid medical conditions.
* Patients who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
* ASA class 4-5.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Successful EGD | Within 24 hours on study day
  Procedure success is assessed at the end of the procedure 1). Procedure success is defined as by successful intubation of the third portion of the duodenum. Photograph of the third portion of the duodenum will be taken.

SECONDARY OUTCOMES:
Endoscopist qualitative rating of the Saneso 360° gastroscope | Within 24 hours on study day
  Endoscopists will rate their experience with the Saneso 360° gastroscope immediately following the completion of the study procedure 1) using a five-point Likert scales (5 - excellent; 4 - good; 3- acceptable; 2- difficult; and 1-unacceptable).
Endoscopist qualitative rating of the Saneso 360° gastroscope compared to their past experience with traditional gastroscopes (TG) | Within 7 days of completion of the study
  Endoscopist qualitative rating of the Saneso 360° gastroscope compared to their past experience with traditional gastroscopes (TG) as it pertains to various design and performance related attributes using a 3-point Likert scale (Saneso gastroscope is 5 - superior to TG; 3 - the same as TG; 1 - inferior to TG).
Evaluation of adverse events (AEs) related to the device. | Within 7 days of completion of the study
  AEs are assessed through 7 days after the procedure.
Evaluation of any potential mucosal injury | Immediately after the use of the device
  Evaluation of any potential mucosal injury resulting from use of the study device immediately following the use of the device (0- no mucosal damage; 1- erythema; 2-bleeding; 3- superficial mucosal tear; 4- deep mucosal tear).

CONTACTS AND LOCATIONS:
Overall Officials: George Goetz, M.D; Ph.D., Principal Investigator — West Virginia School of Medicine, Morgantown, WV
Locations (6):
- United States (6):
  - Valley Endoscopy Center, Saint Clairsville, Ohio
  - Wintersville Endoscopy Center, Wintersville, Wintersville, Ohio
  - West Virginia University School of Medicine - Davis Medical Center, Elkins, West Virginia
  - West Virginia University School of Medicine - Reynolds Memorial Hospital, Glendale, West Virginia
  - West Virginia University School of Medicine - Reynolds Memorial Hospital,, Glendale, West Virginia
  - West Virginia University School of Medicine - Wheeling Hospital, Wheeling, West Virginia

IPD SHARING:
Plan to Share IPD: No